CLINICAL TRIAL: NCT03543150
Title: Botox Drug Use Investigation (Spasmodic Dysphonia)
Brief Title: BOTOX® Drug Use Investigation (Spasmodic Dysphonia)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 208506
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Dysphonia
Keywords: Spasmodic Dysphonia; VHI-10 scores; BOTOX; Drug use investigation
MeSH Terms: conditions — Dysphonia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects receiving BOTOX: Subjects with a diagnosis of spasmodic dysphonia, for which BOTOX is indicated, will be included.
  Interventions: Drug: BOTOX

INTERVENTIONS:
Drug: BOTOX — BOTOX injections will be administered to eligible subjects with diagnosis of spasmodic dysphonia. Dose unit, daily dose frequency, date of administration will be at the investigator discretion.

SUMMARY:
This study is a drug use investigation program of BOTOX. The objective of this investigation is to collect and assess information on the safety and efficacy of BOTOX injections in subjects with a diagnosis of spasmodic dysphonia in daily clinical practice. All subjects treated with BOTOX for spasmodic dysphonia after obtaining approval for the indication of BOTOX for spasmodic dysphonia will be included in this study. Approximately 400 subjects will be included in the study. The observation period per subject will be up to 12 months from the date of the first administration of BOTOX. The total study duration will be will be approximately 3 years from the date of approval for the indication of BOTOX for spasmodic dysphonia. BOTOX is a registered trademark of Allergan, Inc.

ELIGIBILITY:
Inclusion Criteria:

* All subjects treated with Botox for spasmodic dysphonia after obtaining approval for the indication of BOTOX for spasmodic dysphonia are included in this study.

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects receiving BOTOX for spasmodic dysphonia after obtaining approval for the indication of BOTOX for spasmodic dysphonia will be included in this study.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-07-20 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse drug reactions | Up to 1 year
  The investigator will collect the information about all adverse drug reactions including diseases and symptoms, occurring after the first administration of Botox, regardless of whether they are related to BOTOX.
Change from Baseline in voice handicap index (VHI)-10 scores | Baseline and up to 1 year
  The VHI is a 30-item questionnaire divided into 3 subsections including functional, physical, and emotional which measures the effect of voice problems on quality of life. Subjects will mark each item on this 30-item questionnaire on a scale ranging from 0-4 (0 being never and 4 being always). Points for each subscale are tallied and a total composite score is also given. A total score of 0-11 is considered normal, 12-28 is considered mild minimal handicap, 29-56 is considered moderate handicap, and 57-120 is considered severe handicap.
Efficacy rate based on global assessment of efficacy | Up to 1 year
  The efficacy rate is the number of subjects assessed as "effective" based on the course of subjective symptoms and clinical symptoms during the observation period from the date of the first administration of BOTOX injections.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Iimura S, Nose Y, Tabata K, Oda K, Yamashita Y, Takahashi N, Kawano Y. Safety and Effectiveness of OnabotulinumtoxinA in Patients with Laryngeal Dystonia: Final Report of a 52-Week, Multicenter Postmarketing Surveillance Study. Toxins (Basel). 2023 Sep 5;15(9):553. doi: 10.3390/toxins15090553. PMID 37755979